CLINICAL TRIAL: NCT02726490
Title: Glyburide vs Glucovance in the Treatment of Gestational Diabetes
Brief Title: Glyburide vs Glucovance in the Treatment of GDM
Acronym: GGIG
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of Recruitment
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E16008
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes, pregnancy, diabetes
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus | interventions — Glyburide; Glucovance; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glyburide (Active Comparator): * Patients will check and record blood glucose fasting and 1 hour after each meal each day. Patients will also keep a diary of all meals.
  * The starting dose of glyburide may be 2.5milligrams (mg) to 5mg every day(QD) or twice daily (BID) depending on the degree of hyperglycemia.
  * The dose of glyburide will be increased as needed to a maximum of 20mg /day.
  * Antenatal testing will be initiated at 28 weeks
  * Patients will receive monthly growth scans
  Interventions: Drug: Glyburide
- Glucovance (Active Comparator): * Patients will check and record blood glucose fasting and 1 hour after each meal each day. Patients will also keep a diary of all meals.
  * The starting dose of glucovance may be 1.25/250milligrams (mg) either once daily (QD) or twice a day (BID) increased to a maximum of 20mg/2000mg as needed.
  * Patients will receive monthly growth scans
  * Antenatal testing will be initiated at 28 weeks.
  Interventions: Drug: Glucovance

INTERVENTIONS:
Drug: Glyburide — glyburide 2.5milligrams (mg) at bedtime (qhs) increased as needed to a maximum of 20mg/day usually taken twice a day (BID)
  Other Names: micronase; diabeta; glynase
  Arms: Glyburide
Drug: Glucovance — glucovance (2.5/500) 1 taken orally (PO) at bed time (QHS) increased as needed to a maximum dose of (20/2000)/day usually taken twice a day (BID)
  Other Names: combination glyburide and metformin
  Arms: Glucovance

SUMMARY:
A randomized comparison of glyburide to glucovance (metformin -glyburide) in the management of diabetes in pregnancy.

DETAILED DESCRIPTION:
This study will be a randomized open label trial of glyburide compared to glucovance in the management of gestational diabetes. We hypothesize that glucovance will provide improved glycemic control and a lower failure rate with no increase in neonatal adverse outcomes. Sixty-seven patients will be randomized by computer to each arm of the study. Outcomes will be glycemic control, failure rate of the drug to achieve glycemic goals, and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Gestational diabetes
* Pregnancy > 12 weeks gestation
* Ability to give consent

Exclusion Criteria:

* Inability to consent to the study
* Pre-existing diabetes
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Serum creatinine >1
* Liver disease
* Allergy to sulfa;
* Allergy to glyburide;
* Allergy to metformin;
* Fetal anomalies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-07; Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
efficacy of glyburide compared to glucovance | during the index pregnancy
  failure rate of glyburide compared to glucovance in ability to achieve euglycemia

SECONDARY OUTCOMES:
maternal hypoglycemia | during the index pregnancy
  the rate of maternal hypoglycemia associated with each drug
neonatal birthweight | at birth
  infant weight at birth
neonatal apgar scores | at birth
  infant 1 minute and 5 minute apgar scores
neonatal admission to the newborn intensive care unit (NICU) | at birth or within the first 24 hours after birth
  admission to the Newborn intensive care unit (NICU)
neonatal hypoglycemia | up to 24 hours after delivery
  failure of the neonate to maintain blood glucose > 60 milligrams/deciliter (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa E Moore, MD, Principal Investigator — Texas Tech Health Sciences Center El Paso
Locations (1):
- TTUHSC El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore LE, Briery CM, Clokey D, Martin RW, Williford NJ, Bofill JA, Morrison JC. Metformin and insulin in the management of gestational diabetes mellitus: preliminary results of a comparison. J Reprod Med. 2007 Nov;52(11):1011-5. PMID 18161398
- [Result] Moore LE, Clokey D, Rappaport VJ, Curet LB. Metformin compared with glyburide in gestational diabetes: a randomized controlled trial. Obstet Gynecol. 2010 Jan;115(1):55-59. doi: 10.1097/AOG.0b013e3181c52132. PMID 20027034

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT02726490/Prot_SAP_000.pdf